CLINICAL TRIAL: NCT04663620
Title: Design, Implementation and Assessment of a Comprehensive Community Neonatal Heath Package Utilising Medical and Social Interventions
Brief Title: Saving Babies Lives
Acronym: SBL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HCR17009
Record Dates: First submitted 2020-11-12; First posted 2020-12-11 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Perinatal Mortality
MeSH Terms: conditions — Perinatal Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saving Babies Lives Programme (Active Comparator): Comprehensive neonatal healthcare package
  Interventions: Behavioral: Saving Babies Lives Programme
- No Saving Babies Lives Programme (Placebo Comparator): Control arm
  Interventions: Behavioral: No Saving Babies Lives Programme

INTERVENTIONS:
Behavioral: Saving Babies Lives Programme — Comprehensive neonatal healthcare package
  Arms: Saving Babies Lives Programme
Behavioral: No Saving Babies Lives Programme — No comprehensive neonatal healthcare package
  Arms: No Saving Babies Lives Programme

SUMMARY:
The central hypothesis of this study is that a neonatal healthcare programme that has a significant impact on neonatal mortality and which spans the healthcare journey from village to referral hospital can be developed and implemented in a low-resource rural setting.

This study is a five-year cluster-randomised trial, covering a rural and isolated province in North-Eastern Cambodia. The intervention of this study is the Saving Babies' Lives programme, which is a comprehensive, contextual and iterative neonatal healthcare package. The Saving Babies' Lives programme comprises a training programme for primary care facilities, and participatory action research with community health workers (known in Cambodia as village health support group volunteers). The control is no intervention; standard government service continues. Qualitative and quantitative data collection supports improvements in the iterative programme, and evaluation of the study, with the intention of creating a scalable blueprint.

Wellcome Trust grant number 220211.

DETAILED DESCRIPTION:
Globally the proportion of childhood deaths that occur in the neonatal period is increasing. Since 1990 there has been a 47% reduction in deaths in children less than five years of age. However, this rate of reduction has not been seen in infants four weeks of age or younger (neonates). The reasons why the fall in neonatal mortality has not mirrored that seen in children mortality, is complex and one that is not well explored in the literature. One proposed explanation is that interventions that have been successfully employed to reduce childhood death do not reach the community and it is in the community where most neonates die. Another pervasive perceived barrier to providing neonatal care, particularly in remote and rural areas, is the misconception that neonatal care is difficult and expensive.

Many health problems are rooted in powerlessness. Health education that involves community involvement: dialogue and problem solving, rather than just message giving, is more empowering. Addressing social needs and empowering communities to make decisions about health care needs allows for the design of programmes that account for local practices and beliefs. Up to two-thirds of neonatal deaths could be prevented if neonates were given proper care during and immediately after birth, because the majority of neonatal deaths occur around the time of delivery. Training primary level health care workers to deal with emergency situations that occur around the time of delivery, has been shown to decrease maternal mortality and neonatal mortality It is reported that 79% of deliveries in Cambodia occur in healthcare facilities. The majority of these will occur at primary care facilities. Babies born in primary care facilities who require further care are transferred to the referral hospital. The majority of referral hospitals in Cambodia do not have the resources or skills to effectively deal with neonatal complications for babies born either in health centres or in their on-site maternity wards.

The central hypothesis of this study is that a neonatal healthcare programme that has a significant impact on neonatal mortality and which spans the healthcare journey from village to referral hospital can be developed and implemented in a low-resource rural setting.

This study is a five-year cluster-randomised trial, covering the whole of Preah Vihear province in North-Eastern Cambodia, which is a rural and isolated province. A cluster is defined as a primary care administrative group, as recognised by the provincial health department, and includes all primary care facilities, primary care workers, community health workers, villagers and villages in that geographical area. The study area is divided into 21 clusters. Clusters were pre-assigned to one of two arms: intervention and control. A pilot sequence has only four clusters, to incorporate a pilot phase into study design.

The intervention of this study is the Saving Babies' Lives programme which is a comprehensive, contextual and adaptive neonatal healthcare package. The Saving Babies' Lives Programme will be developed in partnership with the Kingdom of Cambodia Ministry of Health. The programme will be approved by the Ministry of Health and a memorandum of understanding signed with the provincial health director of Preah Vihear province. The control is no intervention; standard government service continues.

The primary care facility intervention component of the Saving Babies' Lives programme involves course-based training combined with continuous in-situ mentoring to support doctors, nurses and midwives and other health worker cadres to improve their practical daily skills in emergency and clinical neonatal care. Essential equipment will be identified and included in the package.

Meetings attended by community health workers (two from each of the villages) will be held to identify problems and concerns around neonatal health care in their own village. Monthly meetings will take place for the group to discuss problems, attempt to arrive at solutions, and share learning. These meetings will be facilitated by the study team who will use participatory action research methodology to: identify problems with provision of, and barriers to seeking, neonatal health care; develop interventions to improve care; implement these interventions; assess the group's perception of the effectiveness of interventions.

A neonatal healthcare assessment tool will be developed that is quantitative and qualitative in nature. It will be based on the 'KAP' survey method of analysing Knowledge, Attitudes and Practice. In addition, two further domains will be added, equipment and staffing, leading to a 'KAPES' model of assessment.

Data will be collected and used to assess the impact of the programme, its perceived facilitators and barriers and its successes and failures. This information will be used to iterate the programme content and structure in order to improve it, with the intention of creating a scalable blueprint.

ELIGIBILITY:
Saving Babies Lives Training Programme

Study Participants

The Saving Babies Lives Programme will be aimed at government health care staff working in the community (Village Health Support Group Workers, (VHSG)), at Health Center (nurses and midwives) and at the referral hospital (doctors and nurses)

Inclusion Criteria

• Staff members chosen by the Provincial Health Director to attend the programme

Exclusion Criteria

• Not applicable

Village Health Support Group Workers (VHSG) Baby Health Meetings

Study Participants

* Two Village Health Support Group Workers (VHSG) from villages served by each Health Center cluster
* Adults (aged 18 years or older)

Inclusion Criteria

* Work as a government health care staff working in the community (Village Health Support Group Workers , (VHSG))
* Live in a village served by a chosen Health Center
* Are able to commit to attend meetings regularly
* Give consent to participate in the meetings

Exclusion Criteria

* Refusal to participate
* Be from a village where two members have already been chosen

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24040 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
1. Number of new locations the Saving Babies' Lives programme is replicated in, as assessed by implementation of the programme in a new location | 5 years
  'New location' is defined as consisting of at least one government-run primary care facility (and it's affiliated primary care workers and community health workers) in Cambodia that has not had the Saving Babies' Lives programme implemented before

SECONDARY OUTCOMES:
Change in perinatal mortality rate as assessed using a surveillance system in Preah Vihear province | 5 years

OTHER OUTCOMES:
Causes of death (cause-specific mortality fraction) of all stillbirths and neonates that die as assessed using a verbal autopsy tool | 5 years
Change in neonatal mortality rate as assessed using a surveillance system in Preah Vihear province | 5 years
Percentage of correct knowledge as assessed using a bespoke Knowledge, Attitudes, Practice, Equipment, Staffing annual survey for primary care facilities, change in intervention clusters compared to control clusters | 5 years
Percentage of positive attitudes towards neonatal care as assessed using a bespoke Knowledge, Attitudes, Practice, Equipment, Staffing survey for primary care facilities, change in intervention clusters compared to control clusters | 5 years
Percentage of correct practice as assessed using a bespoke Knowledge, Attitudes, Practice, Equipment, Staffing survey for primary care facilities, change in intervention clusters compared to control clusters | 5 years
Percentage of correct equipment available as assessed using a bespoke Knowledge, Attitudes, Practice, Equipment, Staffing survey for primary care facilities, change in intervention clusters compared to control clusters | 5 years
Percentage of correct staffing practice as assessed using a bespoke Knowledge, Attitudes, Practice, Equipment, Staffing survey for primary care facilities, change in intervention clusters compared to control clusters | 5 years
Satisfaction scores of primary facility workers as assessed by a 5-point likert scale using participant feedback surveys at the end of the training | 5 years
Attendance rates of primary care workers to the training programme as assessed using attendance register records | 5 years
Percentage of correct knowledge as assessed using a bespoke Knowledge, Attitudes, Practice annual survey for community health workers, change in intervention clusters compared to control clusters | 5 years
Percentage of positive attitudes towards neonatal care as assessed using a bespoke Knowledge, Attitudes, Practice survey for community health workers, change in intervention clusters compared to control clusters | 5 years
Percentage of correct practice as assessed using a bespoke Knowledge, Attitudes, Practice survey for community health workers, change in intervention clusters compared to control clusters | 5 years
Satisfaction scores of community health workers as assessed by a 5-point likert scale using participant feedback surveys at the end of the participatory action research | 5 years
Attendance rates of community health workers to the monthly participatory action research meetings as assessed using attendance register records | 5 years
Number of changes to official documentation (policy, strategy, guidelines, training materials) made by the Cambodian Ministry of Health based on the Saving Babies Lives programme as assessed by reviewing all available relevant documents at study end | 5 years
Disability-adjusted life years averted as assessed by cost analysis of the intervention compared to normal standard of care at study end | 5 years
Quality-adjusted life years gained as assessed by cost analysis of the intervention compared to normal standard of care at study end | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Angkor Hospital for Children, Siem Reap, Cambodia

IPD SHARING:
Plan to Share IPD: Yes
Data collected for this study will be under the custodianship of AHC, will be de-identified and may be shared with other groups of researchers in accordance with the current MORU Data Sharing Policy. All applications will be carefully reviewed by the MORU Data Access Committee before granting any approvals to access data. All researchers accessing the data need to adhere to a set of terms and conditions that aim to protect the interests of research participants and other relevant stakeholders.
URL: https://angkorhospital.shinyapps.io/SBLP/

REFERENCES:
- [Derived] Patel K, Say S, Leng D, Prak M, Lo K, Mukaka M, Riedel A, Turner C. Saving babies' lives (SBL) - a programme to reduce neonatal mortality in rural Cambodia: study protocol for a stepped-wedge cluster-randomised trial. BMC Pediatr. 2021 Sep 7;21(1):390. doi: 10.1186/s12887-021-02833-7. PMID 34493225

DOCUMENTS (2):
  • Study Protocol (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/20/NCT04663620/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT04663620/SAP_001.pdf